CLINICAL TRIAL: NCT05371132
Title: Pilot Phase I Study to Evaluate CD8 PET Imaging as a Marker of Immune Response to Stereotactic Body Radiation Therapy (ELIXR)
Brief Title: Study to Evaluate CD8 PET Imaging as a Marker of Immune Response to Stereotactic Body Radiation Therapy (ELIXR)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21221; NCI-2022-02037 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21221 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2022-03-24; First posted 2022-05-12 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Malignant Solid Neoplasm; Lymphoma
MeSH Terms: conditions — Neoplasm Metastasis; Lymphoma | interventions — Magnetic Resonance Spectroscopy; Radiosurgery; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Basic science (zirconium Zr 89-Df-crefmirlimab, PET, SBRT) (Experimental): Patients receive zirconium Zr 89-Df-crefmirlimab IV over 5-10 minutes and then under PET imaging 24 hours after infusion before and after SBRT. Patients undergo SBRT every 2-5 days for a total of 5 fractions. For lymphoma patients only, IMRT on consecutive days may be used.
  Interventions: Procedure: Positron Emission Tomography; Radiation: Stereotactic Body Radiation Therapy; Drug: Zirconium Zr 89-Df-Crefmirlimab; Radiation: Intensity Modulated Radiation Therapy

INTERVENTIONS:
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
Drug: Zirconium Zr 89-Df-Crefmirlimab — Given IV
  Other Names: 89Zr-Crefmirlimab Berdoxam; 89Zr-Desferrioxamine-IAB22M2C; 89Zr-Df-Crefmirlimab; 89Zr-Df-IAB22M2C; Zirconium Zr 89-Df-IAB22M2C; ZIRCONIUM ZR-89-DESFERRIOXAMINE-IAB22M2C
Radiation: Intensity Modulated Radiation Therapy — IMRT for Lymphoma patients only
  Other Names: IMRT

SUMMARY:
"This phase I trial investigates the effect of radiation therapy on the immune system, specifically CD8 positive (+) T cells, in lymphoma patients receiving bridging radiation therapy before CAR T-cell infusion, and metastatic patients with solid tumor malignancies receiving SBRT. CD8+ T cells are mainly found in lymph tissue and play a significant role in anti-tumor immunity. These cells can infiltrate tumor cells and kill them. Radiation therapy may recruit CD8 T cells and this recruitment may help with tumor control. Diagnostic procedures, such as zirconium Zr 89-Df-crefmirlimab positron emission tomography (PET), may be a less invasive way to check and monitor for CD8+ T cells before and after radiation therapy."

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate if there is an increase in CD8+ T cells after stereotactic body radiation therapy (SBRT) in irradiated tumors.

SECONDARY OBJECTIVES:

I. To report on the time evolution of zirconium Zr 89-Df-crefmirlimab (CD8 PET tracer) uptake after infusion.

II. To compare CD8 PET tracer uptake at irradiated lesions to uptake at non-irradiated lesions (if any).

III. To assess how differences in site, histology and/or prior therapy relate to immune characterization and changes IV. To assess serum biomarkers of immune response before and after SBRT. V. To assess ability of CD8 PET tracer and imaging to be a biomarker of SBRT. VI. Evaluate CD8 PET tracer with Response Evaluation Criteria in Solid Tumors (RECIST) radiology measurements.

VII. To report any adverse events associated with 2 doses of CD8 PET tracer when used in combination with SBRT.

EXPLORATORY OBJECTIVE:

I. Blood will be collected, processed, and stored for future immune profiling or other correlatives pending additional funding.

II. Evaluate the safety and feasibility of using CD8 PET imaging to assess immune system activation during and after bRT for CAR T cell therapy.

III. Describe the CD8 PET tracer uptake prior to CAR T and the response/duration of response to CAR T cell therapy

OUTLINE:

Patients receive zirconium Zr 89-Df-crefmirlimab intravenously (IV) over 5-10 minutes and then undergo PET imaging 24 hours after infusion before and after SBRT. Patients undergo SBRT every 2-5 days for a total of 5 fractions.

The subset of lymphoma patients enrolled on trial who are being treated in the bridging radiation setting before CAR T-cell therapy will receive 3 infusions of Zr89-Df-crefmirlimab and associated CD8 ImmunoPET imaging before radiation, after radiation, and after CAR T-cell infusion.

After completion of study treatment, patients are followed up at 4-6 weeks, 3 months, 1 year, and then periodically for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Participant is willing and able to comply with all protocol required procedures
* Age: >= 18 years
* Eastern Cooperative Oncology Group (ECOG) =< 2
* Metastatic patients of any solid tumor malignancy amenable for SBRT as determined by the radiation oncologist
* Lymphoma patients may be allowed as determined by the principal investigator (PI)
* No change in systemic treatment regimen for past 2 months prior to start of SBRT
* Patients able to comply with daily PET after SBRT
* Patient meets all clinical safety lab values per institution's standard of care, or Investigator's discretion, for patients receiving cancer treatment
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use effective double barrier contraceptive methods or abstain from heterosexual activity for the course of the study through at least 30 days after the last administration of the CD8 PET tracer

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Patient who have splenic disorders or had splenectomy that per PI would interfere with CD8 imaging
* Patients should not have any uncontrolled illness including ongoing or active infection
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CD8 PET tracer
* Serious nonmalignant disease or conditions that could compromise protocol objectives, in the opinion of the investigator
* Females only: Pregnant or breastfeeding

  * Pregnant women are excluded from this study because CD8 PET tracer is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with CD8 PET tracer, breastfeeding should be discontinued if the mother is treated with CD8 PET tracer
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2026-10-05 (Estimated); Study Completion 2026-10-05 (Estimated)

PRIMARY OUTCOMES:
Change in CD8 positron emission tomography (PET) maximum standardized uptake value (SUVmax) | Pre-SBRT to post-SBRT (comparison of CD8 PET SUV at day -1, and at 1 week after completion of SBRT)
  CD8 PET SUV will be measured as SUVmax, the maximum SUV measurement within the tumor voxels. If patients have multiple tumors treated with stereotactic body radiation therapy (SBRT), average within-tumor change will be used for that patient for the primary analysis. As a result, this primary analysis is a comparison of the change in CD8 PET SUV in 10 patients.

SECONDARY OUTCOMES:
Time evolution of CD8 PET SUV (decay corrected) | From pre-SBRT to post-SBRT (comparison of CD8 PET SUV at day -1, and at each of 5 fractions of SBRT administered 2-5 days apart, and additional imaging 1-2 weeks after completion of SBRT)
  CD8 PET SUVs from PET scans taken before, during and after SBRT.
Site specific differences in immune characterization (CD8 PET SUV) and changes | From pre-SBRT to post-SBRT ( CD8 PET SUV at day -1, and at each of 5 fractions of SBRT administered 2-5 days apart, and additional imaging 1-2 weeks after completion of SBRT).
  CD8 PET SUV and change in CD8 PET SUV at tumor sites will be collected to assess whether immune activity and response is different at different sites of disease (e.g., lymph node vs bone)
Histology specific differences in immune characterization (CD8 PET SUV) and changes | From pre-SBRT to post-SBRT ( CD8 PET SUV at day -1, and at each of 5 fractions of SBRT administered 2-5 days apart, and additional imaging 1-2 weeks after completion of SBRT).
  CD8 PET SUV and change in CD8 PET SUV will be collected to assess whether immune activity and response is different depending on the patient's disease type and histopathology.
Evaluation of tumor response (fludeoxyglucose F-18 [FDG] PET and/or computed tomography [CT]) as it relates to both baseline CD8 PET SUV and changes observed after SBRT. | Pre-SBRT to post-SBRT (1-2 weeks after completion of SBRT). Additional RECIST response assessments will be conducted per standard of care and will be assessed for up to 2 years to compare to CD8 SUVs post-SBRT and changes in CD8 SUVs.
  RECIST response and evaluation endpoints will be used to assess tumor response from CT imaging, and SUVmax will be used for FDG-PET imaging. Data will be compared with CD8 PET SUVs (e.g. SUVmax of CD8 PET) and changes pre- and post-SBRT. For multiple lesions irradiated SUVmax will be averaged.
CD8 PET SUV (Subset) | Pre-bridging radiation to post-CAR T cell therapy (approximately at least 7 days after CAR T cell infusion). Additional response and survival data will be collected up to 2 years after completion of study therapy.
  Will describe CD8 PET SUV in the subset (approximately 2 patients) who receive CAR-T therapy, and those patients' response/duration of response to CAR-T. CD8 PET SUVs from PET scans taken before, during and after bridging radiation, as well as after CAR T cell therapy. Response to radiation and CAR T and survival after the combination treatment will be collected and compared to CD8 uptake patterns.
Incidence of adverse events | From the first CD8 PET tracer infusion to 4-6 weeks after the last CD8 PET tracer infusion.
  Number and type of adverse events related to the study treatment

OTHER OUTCOMES:
Correlation between immune characterization of blood samples and CD8 PET SUVs and tumor response | Pre-SBRT to post-SBRT (1 week after completion of SBRT)
  Changes in circulating levels of immune cells and cytokines will be compared to changes in CD8 PET SUVs and tumor response (measured by RECIST or FDG PET SUVs). If multiple lesions, the average will be used. Most metrics will use SUVmax, although others will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Savita V Dandapani, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States